CLINICAL TRIAL: NCT00549419
Title: Randomized Evaluation of Arterial Pressure Based Cardiac Output for Goal-Directed Therapy in Patients Undergoing Major Abdominal Surgery
Brief Title: Arterial Pressure Based Cardiac Output for Goal-Directed Therapy in Abdominal Surgery
Acronym: REPEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinikum Ludwigshafen (Other)
Responsible Party: Stefan Suttner, Klinikum Ludwigshafen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-06
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-01

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Ringer's Lactate; Hydroxyethyl Starch Derivatives; Norepinephrine; Dobutamine; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In the Treatment group, the traditional vital signs and APCO are made continuously available for fluid and catecholamine optimization and clinical decision making.
  Interventions: Drug: Goal-directed hemodynamic therapy
- 2 (Active Comparator)
  Interventions: Drug: Ringers lactate, hydroxyethyl starch; norepinephrine, dobutamine; Drug: Standard of care

INTERVENTIONS:
Drug: Ringers lactate, hydroxyethyl starch; norepinephrine, dobutamine — The Control group will be assessed using the standard care of traditional vital signs
  Arms: 2
Drug: Goal-directed hemodynamic therapy — Ringers lactate, hydroxyethyl starch; norepinephrine, dobutamine
  Arms: 1
Drug: Standard of care — Ringers lactate, hydroxyethyl starch; norepinephrine, dobutamine
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the early identification and more precise intervention of goal-directed intraoperative plasma volume expansion and catecholamine therapy using arterial pressure based cardiac output (APCO) measurement in addition to normal vital signs will improve postoperative organ function, in particular renal function, in patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for elective major abdominal surgery and has two or more risk factors according to the Lee classification scheme.
* Patient can sign informed consent before surgery.
* Patient is able to comply with the study procedure.
* Patient must require an indwelling radial or a femoral artery catheter.
* Patient must be 20 years old or older.
* Patient must be 40kg or heavier.
* Patients height and weight can be accurately obtained prior to study start.

Exclusion Criteria:

* Emergency surgery.
* Patients with aortic or mitral valve regurgitation.
* Renal insufficiency requiring hemodialysis.
* Liver dysfunction (alanine/aspartate aminotransferase >40 U/L).
* Patient with contraindications for the placement of radial, femoral or other arterial cannulae.
* Patient being treated with an intraaortic balloon pump.
* Female patients with a known pregnancy.
* Patient is currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is postoperative renal function, as determined by measurement of the glomerular filtration rate. | 6 month

SECONDARY OUTCOMES:
Total fluid requirements (type and volume); Drug requirement (type and volume); Other organ function (myocardial function, liver function, endothelial function, degree of inflammation) | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan W. Suttner, M.D. Ph.D., Study Director — Klinikum Ludwigshafen
Locations (1):
- Klinikum Ludwigshafen, Ludwigshafen, RLP, Germany

REFERENCES:
- [Derived] Mayer J, Boldt J, Mengistu AM, Rohm KD, Suttner S. Goal-directed intraoperative therapy based on autocalibrated arterial pressure waveform analysis reduces hospital stay in high-risk surgical patients: a randomized, controlled trial. Crit Care. 2010;14(1):R18. doi: 10.1186/cc8875. Epub 2010 Feb 15. PMID 20156348